CLINICAL TRIAL: NCT01139138
Title: A Phase IB/II Study of Second Line Therapy With Panitumumab, Irinotecan and Everolimus (PIE) in Metastatic Colorectal Cancer With KRAS WT
Brief Title: Safety Study of the Combination of Panitumumab, Irinotecan and Everolimus in the Treatment of Advanced Colorectal Cancer
Acronym: PIE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Queen Elizabeth Hospital (Other)
Collaborators: Amgen (Industry); Novartis (Industry)
Responsible Party: Principal Investigator, Amanda Townsend, Dr, The Queen Elizabeth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AU-2009-0003/CRAD001CAU06T
Record Dates: First submitted 2010-05-28; First posted 2010-06-08 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumors; Neoplasms, Colorectal
Keywords: Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumors; Neoplasms, Colorectal
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Irinotecan; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab + Irinotecan + Everolimus (Experimental)
  Interventions: Drug: Panitumumab; Drug: Irinotecan; Drug: Everolimus

INTERVENTIONS:
Drug: Panitumumab — Panitumumab 6mg/kg IV every 14 days
  Other Names: Vectibix
Drug: Irinotecan — Irinotecan 200mg/m2 IV every 14 days
Drug: Everolimus — Everolimus daily po (dosage varies with cohort)
  Other Names: RAD001

SUMMARY:
This study will assess the safety of panitumumab, irinotecan and everolimus when given in combination to treat advanced colorectal cancer

DETAILED DESCRIPTION:
This is an open label uncontrolled phase IB/II study to determine the maximum tolerated dose (MTD) and assess the efficacy of everolimus, irinotecan and panitumumab when given in combination for patients with metastatic colorectal cancer and KRAS wild-type (WT). Patients with metastatic colorectal cancer (mCRC) that have failed fluorouracil based first line therapy will be included. It is anticipated that approximately 50 patients will be enrolled over a period of 24 months

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histological diagnosis of colorectal cancer that is KRAS wild type
* Metastatic disease not amenable to resection
* Measurable disease as assessed by CT scan using RECIST criteria
* Received and failed fluoropyrimidine therapy
* Radiographically documented disease progression per RECIST criteria
* For phase 1b group only, ECOG PS 0-1
* For phase 2 group only, ECOG PS 0-2
* Adequate bone marrow function with haemoglobin > 100 g/L, platelets > 100 X 109/l; neutrophils > 1.5 X 109/l within 7 days of enrolment
* Adequate renal function, with calculated creatinine clearance >40 ml/min (Cockcroft and Gault) within 7 days of enrolment
* Adequate hepatic function with serum total bilirubin < 1.25 X upper limit of normal range and ALT or AST<2.5xULN (<5xULN if liver metastases present) within 7 days of enrolment
* Magnesium ≥ lower limit of normal within 7 days of enrolment.
* Fasting serum cholesterol ≤ 7.75mmol/L AND fasting triglycerides ≤ 2.5 x ULN. Note: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Life expectancy of at least 12 weeks
* Negative pregnancy test ≤ 72 hours before commencing study treatment (women of childbearing potential only).
* Written informed consent including consent for biomarker studies

Exclusion Criteria:

* Presence of KRAS mutation in tumour sample
* For Phase 1b group only, patients with prior pelvic radiotherapy.
* Systemic chemotherapy, immunotherapy, approved proteins/antibodies or any investigational agent within 4 weeks prior to commencing study treatment
* Radiotherapy within 14 days of commencing study treatment.
* Unresolved toxicities from prior systemic therapy or radiotherapy
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or to complete the protocol
* Prior treatment with drugs targeting EGFR such as cetuximab, panitumumab or erlotinib
* Prior therapy with mTOR inhibitors (sirolimus, temsirolimus, everolimus)
* Prior therapy with irinotecan
* CYP3A4 enzyme inducing anti-convulsant medication ≤ 14 days prior to study treatment.
* Ketoconazole ≤ 7 days before study treatment.
* Uncontrolled diabetes mellitus defined by fasting glucose >1.5 x ULN.
* Known cirrhosis, chronic active hepatitis, or chronic persistent hepatitis
* Patients with known interstitial lung disease or severely impaired lung function
* Patients with active bleeding diatheses.
* Any uncontrolled clinically significant cardiac disease, arrhythmias or angina pectoris
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhoea
* Chronic treatment with immunosuppressives
* Patients with a known history of HIV seropositivity
* Patients who have any severe and/or uncontrolled medical conditions or infections
* Untreated or symptomatic CNS metastases
* Patients who have a history of another primary malignant disease
* Pregnancy or lactation.
* Women and partners of women of childbearing potential who are not using effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-06; Primary Completion 2015-08 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities | at end of cycle 2 (each cycle is 14 days)
  To determine the maximum tolerated dose (MTD)of everolimus, irinotecan and panitumumab when given in combination for patients with Kras WT mCRC

SECONDARY OUTCOMES:
Safety & toxicity | Approximately 24 weeks
  Safety and toxicity assessed weekly during the phase Ib component (as per NCI CTCAE version 3.0) and fortnightly during the phase II component
Response rate | Assessed every 6 weeks until disease progression
  Objective tumour response as per RECIST criteria V1.0
Progression free survival | Until disease progression, occurrence of new disease or death
Overall Survival | Assessed 3 monthly until death

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Townsend, MBBS, Principal Investigator — The Queen Elizabeth Hospital
Locations (1):
- The Queen Elizabeth Hospital, Adelaide, South Australia, Australia